CLINICAL TRIAL: NCT00003857
Title: Phase III Trial of Tamoxifen Alone vs. Tamoxifen Plus Radiation Therapy for Good Risk Duct Carcinoma In-Situ (DCIS) of the Female Breast
Brief Title: Radiation Therapy With or Without Optional Tamoxifen in Treating Women With Ductal Carcinoma in Situ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9804; CDR0000067020; CAN-NCIC-MA26; CALGB-49801; NCI-2011-02038 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: breast cancer in situ; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Tamoxifen; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation +/- tamoxifen for 5 years (Active Comparator): Observation +/- tamoxifen 20 mg per day for 5 years
  Interventions: Drug: tamoxifen citrate; Procedure: adjuvant therapy
- Radiation therapy +/- tamoxifen for 5 years (Experimental): Radiation therapy to the whole breast +/- tamoxifen 20 mg per day for 5 years
  Interventions: Drug: tamoxifen citrate; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: tamoxifen citrate
Procedure: adjuvant therapy
Radiation: radiation therapy
  Arms: Radiation therapy +/- tamoxifen for 5 years

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen by the tumor cells. It is not yet known if radiation therapy is more effective than observation, with or without tamoxifen, in treating ductal carcinoma in situ.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with that of observation, with or without tamoxifen, in treating women who have ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of whole breast radiotherapy vs observation with or without optional tamoxifen in decreasing or delaying the appearance of local failure (both invasive and in situ) and preventing the need for mastectomy in women with good-risk ductal carcinoma in situ (DCIS) of the breast.
* Compare distant disease-free survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (under 50 vs 50 and over), final path margins (negative vs 3-9 mm vs at least 10 mm), mammographic size of primary (no greater than 1 cm vs greater than 1 cm to 2.5 cm), nuclei grade (low vs intermediate), and tamoxifen use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo observation and may receive optional oral tamoxifen once daily (at the discretion of the physician) for 5 years.
* Arm II: Beginning within 12 weeks after final surgery, patients receive radiotherapy to the whole breast once daily, 5 days a week, for 3.5-5.5 weeks. Patients may receive optional tamoxifen as in arm I.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,790 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Ductal carcinoma in situ (DCIS) of the breast detected by mammogram at the time of diagnosis

  * Unicentric
  * Lesions ≤ 2.5 cm
  * Low nuclei grade (NG1) or intermediate nuclei grade (NG2) with necrosis in < one third of the involved ducts
  * Inked margins ≥ 3 mm
  * Clinically node negative
  * Non-palpable
* No suspicious areas on post-operative mammogram taken within 12 weeks after final surgery
* No bloody nipple discharge
* No more than 12 weeks since prior final surgery (arm II only)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 26 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* No active connective tissue disorders (e.g., lupus or scleroderma)
* No prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No other concurrent hormonal therapy (e.g., raloxifene, hormone replacement therapy, or birth control pills)

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 26 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 1999-12 (Actual); Primary Completion 2004-02 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Local recurrence (e.g., invasive or noninvasive recurrence) | From randomization to date of local failure in the treated breast or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.

SECONDARY OUTCOMES:
Overall survival | From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.
Time to distant metastasis | From randomization to date of distant metastasis or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.
Invasive local recurrence | From randomization to date of invasive local failure in the treated breast or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.
Salvage mastectomy rate | Analysis occurs after all patients have been potentially followed for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Beryl McCormick, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Clifford A. Hudis, MD — Memorial Sloan Kettering Cancer Center; Barbara L. Smith, MD, PhD, Study Chair — Massachusetts General Hospital; Timothy J. Whelan, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre; Eileen Rakovitch, MD — Toronto Sunnybrook Regional Cancer Centre
Locations (369):
- United States (305):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Saint Joseph's Mercy Cancer Center, Hot Springs, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Mount Diablo Regional Cancer Center, Concord, California
  - North Bay Cancer Center, Fairfield, California
  - Washington Township Hospital, Fremont, California
  - Saint Agnes Medical Center, Fresno, California
  - Cancer Care Consultants Medical Associates at Daniel Freeman Memorial Hospital, Inglewood, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Memorial Medical Center Cancer Services, Modesto, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Torrance Memorial Medical Center, Torrance, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Ruby L. Golleher Cancer Program at Presbyterian Intercommunity Hospital, Whittier, California
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Leeward Radiation Oncology Center, ‘Ewa Beach, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Good Shepherd Hospital, Barrington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Cancer Center at St. John's Medical Center, Anderson, Indiana
  - Regional Cancer Institute at Bloomington Hospital, Bloomington, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Treatment Center for Southern Kentucky, Bowling Green, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Medical Center - Bramhall Campus, Portland, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Bethke Cancer Center at Emerson Hospital, Concord, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital, Fall River, Massachusetts
  - MetroWest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Community Cancer Care at Milford Regional Medical Center, Milford, Massachusetts
  - Caritas Norwood Hospital, Norwood, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth - Hitchcock Concord, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth-Douglass Hospital, Dover, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Albuquerque Regional Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Long Island College Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cancer Treatment Center at Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - St. Joseph Cancer Center at St. Joseph Health Center, Warren, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase-Temple Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Wellspan Health, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Columbia St. Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - West Allis Memorial Hospital, West Milwaukee, Wisconsin
- Canada (64):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Lethbridge Cancer Centre, Lethbridge, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Nanaimo Cancer Clinic at Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Providence Health Care - Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Royal Victoria Hospital of Barrie, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchner, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Centre - Mississauga Site, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - North York General Hospital - Ontario, North York, Ontario
  - Male Health Centre - Oakville, Oakville, Ontario
  - R. S. McLaughlin Durham Regional Cancer Centre at Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Algoma Regional Cancer Program at Sault Area Hospital, Sault Ste. Marie, Ontario
  - Scarborough Hospital - General Campus, Scarborough Village, Ontario
  - St. Catharines General Hospital at Niagara Health System, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Male Health Centre - North York, Toronto, Ontario
  - St. Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital - Weston, Weston, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Prince Edward Island Cancer Centre at Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Centre de Sante et de Services Sociaux de Chicoutimi, Chicoutimi, Quebec
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Doctor Leon Richard Oncology Centre, Greenfield Park, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - Hotel-Dieu de Levis, Lévis, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Regional de Rimouski, Québec

REFERENCES:
- [Result] McCormick B, Winter K, Hudis C, Kuerer HM, Rakovitch E, Smith BL, Sneige N, Moughan J, Shah A, Germain I, Hartford AC, Rashtian A, Walker EM, Yuen A, Strom EA, Wilcox JL, Vallow LA, Small W Jr, Pu AT, Kerlin K, White J. RTOG 9804: a prospective randomized trial for good-risk ductal carcinoma in situ comparing radiotherapy with observation. J Clin Oncol. 2015 Mar 1;33(7):709-15. doi: 10.1200/JCO.2014.57.9029. Epub 2015 Jan 20. PMID 25605856
- [Derived] McCormick B, Winter KA, Woodward W, Kuerer HM, Sneige N, Rakovitch E, Smith BL, Germain I, Hartford AC, O'Rourke MA, Walker EM, Strom EA, Hopkins JO, Pierce LJ, Pu AT, Sumida KNM, Vesprini D, Moughan J, White JR. Randomized Phase III Trial Evaluating Radiation Following Surgical Excision for Good-Risk Ductal Carcinoma In Situ: Long-Term Report From NRG Oncology/RTOG 9804. J Clin Oncol. 2021 Nov 10;39(32):3574-3582. doi: 10.1200/JCO.21.01083. Epub 2021 Aug 18. PMID 34406870
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/